CLINICAL TRIAL: NCT06434974
Title: Prevalence of Birth Before Arrival and Associated Factors Among Postpartum Women in Southern Ethiopia: Community-Based Cross-Sectional Study
Brief Title: Prevalence of Birth Before Arrival and Associated Factors Among Postpartum Women in Southern Ethiopia
Status: Completed | Type: Observational
Sponsor: Wachemo University (Other)
Responsible Party: Principal Investigator, Mitiku Desalegn, Lecturer, Wachemo University
Other Study IDs: LMHB
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Safe Delivery of Baby
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Interviewer administered questionnaire

SUMMARY:
Background: Birth before arrival is defined as unplanned deliveries without the attendance of skilled personnel just before arrival to a health facility. It constitutes a high-risk newborn population and has high perinatal morbidity and mortality. In Ethiopia, most studies and health surveys done, only look at home and hospital deliveries but do not consider deliveries taking place between the house and health facility. The aim of this study is to assess the prevalence of birth before arrival and its associated factors among postpartum women in Lemo woreda, Hadiya zone, SNNPR Ethiopia, 2023.

Methods: Community-based cross-sectional study was conducted among postpartum women in Lemo woreda, Hadiya zone, SNNPR Ethiopia from April, 05 to May 20, 2023. Three hundred eighty-two postpartum women who gave birth six months preceding this study were included. Twelve out of 36 kebeles were selected randomly and simple random sampling was employed for the selection of participant women. Interviewer-administered questionnaire was used for data collection. A binary logistic regression analysis was computed and variables with a p-value of < 0.25 were recruited to the final multivariable logistic regression analysis. Model fitness was checked using Hosmer and Lemeshow goodness of fit test (x2 = 16.04, p-value = 0.250). Statistical significance was declared using odds ratios and 95% confidence intervals at p-value < 0.05.

Result: The prevalence of birth before arrival among women who gave birth in the last six months preceding this study in the study area was 15.2% (95%CI: 11.8%, 19.1%). In the multi-variable analysis, the variables found to have an association with birth before arrival in the final model were having no antenatal care (AOR = 2.63; 95%CI: 1.23, 5.63), dependent women autonomy status (AOR = 3.32; 95%CI: 1.12, 9.89), being not knowledgeable about labor symptoms (AOR = 2.15; 95%CI: 1.11, 4.18), and having birth preparedness towards index birth (AOR = 0.13; 95%CI: 0.05, 0.35).

Conclusion: The prevalence of birth before arrival in the study area was unacceptably high. A statistically significant association was seen between birth before arrival and having no antenatal care, dependent women's autonomy status, being not knowledgeable about labor symptoms, and having birth preparedness towards index birth. Intervening to avert birth before arrival through effective antenatal care programs and enhancing women's autonomy may help to reduce birth before arrival and its adverse perinatal outcomes.

DETAILED DESCRIPTION:
Results Socio-demographic characteristics A total of 382 study participants were included in the analysis with a 100% response rate. The mean age of participant women was 30.3 years + 4.4 SD. The majority of participant women were in the age group 23-26 years (28.3%), but women in the age category of 27-30 were the most experienced birth before arrival (34.6%) and three fourth of them were rural residents (76.2%). Nearly half of women (45.5%) attained secondary education (grades 9-12). The majority of the participant mothers (83.8%) were housewives in their occupation whereas 68.0% of their husbands were farmers. The mean estimated monthly income of the family was 7,216 birr + 3,073.4 SD. The majority of participants (95.0%) had media exposure and radio was the commonest media (Table 2).

Table 2: Socio-demographic characteristics of women who gave birth in the last six months in Lemo district, Hadiya zone, Southern Ethiopia (n = 382).

Variables Category Frequency (percentage) Total

No BBA BBA Mother's age in years Range (23-38) 23-26 27-30 31-34 35-38 105 (97.2%) 70 (65.4%) 78 (88.6%) 71 (88.9%) 3 (2.8%) 37 (34.6%) 10 (11.4%) 8 (10.1%) 108 (28.3%) 107 (28.0%) 88 (23.0%) 79 (20.7%) Residence Urban Rural 74 (81.3%) 250 (85.9%) 17 (18.7%) 41 (14.1%) 91 (23.8%) 291 (76.2%) Women's educational status No formal education Primary Secondary Higher education 31 (60.8%) 154 (88.5%) 126 (89.4%) 13 (81.3%) 20 (39.2%) 20 (11.5%) 15 (10.6%) 3 (18.7%) 51 (13.4%) 174 (45.5%) 141 (36.9%) 16 (4.2%) Husband's educational status No formal education Primary Secondary Higher education 5 (41.7%) 132 (89.8%) 160 (86.5%) 27 (71.1%) 7 (58.3%) 15 (10.2%) 25 (13.5%) 11 (28.9%) 12 (3.1%) 147 (38.5%) 185 (48.4%) 38 (10.0%) Women's occupation Housewife Maid Civil servant 272 (85.0%) 38 (86.4%) 14 (77.8%) 48 (15.0%) 6 (13.6%) 4 (22.2%) 320 (83.8%) 44 (11.5%) 18 (4.7%) Husband's occupation Farmer Merchant Civil servant 229 (88.1%) 80 (77.7%) 15 (78.9%) 31 (11.9%) 23 (22.3%) 4 (21.1%) 260 (68.0%) 103 (27.0%) 19 (5.0%) Housing characteristics Private Rented 295 (85.3%) 29 (80.6%) 51 (14.7%) 7 (19.4%) 346 (90.6%) 36 (9.4%) The average estimated monthly income of the family in Birr 2,000-6,000 6,001-11,000 11,001-15,000 162 (89.0%) 126 (78.7%) 36 (90.0%) 20 (11.0%) 34 (21.3%) 4 (10.0%) 182 (47.6%) 160 (41.9%) 40 (10.5%) Media exposure Yes No 310 (85.4%) 14 (73.7%) 53 (14.6%) 5 (26.3%) 363 (95.0%) 19 (5.0%) Type of media (n = 363) Radio Television Social media 277 (88.8%) 28 (65.1%) 5 (62.5%) 35 (11.2%) 15 (34.9%) 3 (37.5%) 312 (81.7%) 43 (11.2%) 8 (2.1%) BBA: Birth Before Arrival; birr: Ethiopian currency Reproductive Health and Obstetric Characteristics The majority of participant women (76.7%) of them had antenatal care (ANC) follow-up for their last pregnancy. Two-thirds of women had 1-3 ANC contacts for their last delivery with a mean of 1.2 + 0.4 SD. The proportion of women who used contraceptives before their last pregnancy was 26.4%. Two-thirds of the participant women (71.7%) had postnatal care (PNC) follow-up for their last birth and 76.2% of women had planned and wanted the type of last pregnancy. The average value of the women's autonomy index was 0.68 and 26.7% of participant women were autonomous. The proportion of women with grand multigravida was 21.0%, the duration of labor of index birth > 12 hours was 54.7%, birth preparedness towards index birth of 86.1%, women with knowledge of the expected date of delivery (EDD) of the index birth were 66.7%, and 66.1% of women know labor symptoms. The mean number of pregnancies was 3.0 + 1.6 SD and the median duration of labor of the last birth was 14 (IQR 12-24) (Table 3).

Table 3: Reproductive health and obstetric characteristics of participant women by birth before arrival in Lemo district, Hadiya zone, Southern Ethiopia (n = 382).

Variables Category Frequency (percentage) Total

No BBA BBA ANC for the last delivery Yes No 254 (86.7%) 70 (78.7%) 39 (13.3%) 19 (21.3%) 293 (76.7%) 89 (23.3%) Number of ANC contacts (n = 293) 1-3 contacts > 4 contacts 178 (86.0%) 76 (88.4%) 29 (14.0%) 10 (11.6%) 207 (70.6%) 86 (29.4%) Type of health facility for ANC (n = 293) At hospital At health centre At health post 14 (82.4%) 177 (87.2%) 63 (86.3%) 3 (17.6%) 26 (12.8%) 10 (13.7%) 17 (5.8%) 203 (69.3%) 73 (24.9%) Used contraceptive before last pregnancy Yes No 83 (82.2%) 241 (85.8%) 18 (17.8%) 40 (14.2%) 101 (26.4%) 281 (73.6%) PNC for the last delivery Yes No 233 (85.0%) 91 (84.3%) 41 (15.0%) 17 (15.7%) 274 (71.7%) 108 (28.3%) Type of pregnancy Planned and wanted Unplanned but wanted Unplanned & unwanted 249 (85.6%) 68 (91.9%) 7 (41.2%) 42 (14.4%) 6 (8.1%) 10 (58.8%) 291 (76.2%) 74 (19.4%) 17 (4.4%) Women autonomy Non-autonomous Autonomous 231 (82.5%) 93 (91.2%) 49 (17.5%) 9 (8.8%) 280 (73.3%) 102 (26.7%) Gravidity Multigravidae Grand multigravidae 259 (85.8%) 65 (81.3%) 43 (14.2%) 15 (18.7%) 302 (79.0%) 80 (21.0%) Duration of labor of index birth < 12 hours > 12 hours 155 (89.6%) 169 (80.9%) 18 (10.4%) 40 (19.1%) 173 (45.3%) 209 (54.7%) Know the EDD of the index birth Yes No 226 (88.6%) 98 (77.2%) 29 (11.4%) 29 (22.8%) 255 (66.7%) 127 (33.3%) Birth preparedness towards index birth Yes No 285 (86.6%) 39 (73.6%) 44 (13.4%) 14 (26.4%) 329 (86.1%) 53 (13.9%) Knowledge of labor symptoms (n=350) Not knowledgeable Knowledgeable 89 (74.8%) 205 (88.7%) 30 (25.2%) 26 (11.3%) 119 (34.0%) 231 (66.0%) Mode of previous delivery SVD Instrumental delivery SVD with episiotomy Cesarean section 217 (85.1%) 34 (94.4%) 72 (80.9%) 1 (50.0%) 38 (14.9%) 2 (5.6%) 17 (19.1%)

1 (50.0%) 255 (66.7%) 36 (9.4%) 89 (23.3%) 2 (0.6%) ANC: Antenatal Care; BBA: Birth Before Arrival; EDD: Expected Date of Delivery; PNC: Postnatal Care; SVD: Spontaneous Vaginal Delivery Access to a healthcare facility The median time of the delay to seek health care was 14 hours (IQR 12-24) and the mean duration of the second delay was 1.3 hours + 0.6 SD. One-fourth (25.9%) of women delayed > 24 hours in deciding to seek health care and one-third (33.8%) travelled > 2 hours to reach a health care facility. The major reason for the first delay was not realising the problem (28.8%) for women with birth before arrival and lack of transport (62.3%) was the major reason for the second delay. About means of transport, 35.8% of women used Horse/Donkey carts. Regarding the condition of the road, 29.3% of women replied that it is a wide road. More than half of women (51.6%) delivered their index birth at night (Table 4).

Table 4: Access to health care facility among women who gave birth in the last six months in Lemo district, Hadiya zone, Southern Ethiopia (n=382).

Variables Category Frequency (percentage) Total

No BBA BBA First delay Delayed < 24 hours Delayed > 24 hours 246 (86.9%) 78 (78.8%) 37 (13.1%) 21 (21.2%) 283 (74.1%) 99 (25.9%) Second delay (n = 317) Traveled < 2 hours Traveled > 2 hours 171 (81.4%) 88 (82.2%) 39 (18.6%) 19 (17.8%) 210 (66.2%) 107 (33.8%) Reasons for 1st delay Underestimate severity Did not realize the problem Essential person for decision making not around 195 (86.7%) 116 (71.2%) 78 (86.7%) 30 (13.3%) 47 (28.8%) 12 (13.3%) 225 (100%) 163 (100%) 90 (100%) Reasons for 2nd delay (n = 317) Lack of money Lack of transport Distant health facility 61 (87.1%) 159 (80.7%) 38 (77.6%) 9 (12.9%) 38 (19.3%) 11 (22.4%) 70 (22.1%) 197 (62.3%) 49 (15.6%) Means of transport (n = 317) Motorbike Ambulance Public transport Horse/Donkey cart On foot Carried by other people 39 (100.0%) 16 (48.5%) 62 (100.0%) 83 (73.5%) 14 (58.3%) 44 (97.8%) 0 (0.0%) 17 (51.5%) 0 (0.0%) 30 (26.5%) 10 (41.3%)

1 (2.2%) 39 (12.3%) 33 (10.4%) 62 (19.6%) 113 (35.8%) 24 (7.6%) 45 (14.2%) Status of the roadroad All weather road Weather raod 225 (83.3%) 99 (88.4%) 45 (16.7%) 13 (11.6%) 270 (70.7%) 112 (29.3%) Time of delivery of index birth Night Day 150 (76.1%) 174 (94.1%) 47 (23.9%) 11 (5.9%) 197 (51.6%) 185 (48.4%) Women who delivered their last birth at home were not asked for the second delay and its reasons.

Birth before arrival The prevalence of birth before arrival among women who gave birth in the last six months preceding this study in the study area was 15.2% (95%CI: 11.8%, 19.1%). Among them, 84.5% of women gave birth on the route to a health care facility (Table 5).

Table 5: Profile of birth before arrival among women who gave birth in the last six months in Lemo district, Hadiya zone, Southern Ethiopia (n = 382).

Variables Frequency Percentage Place of last delivery Home Before arrival to a health care facility Health care facility 67 58 257 17.5 15.2 67.3 The specific place of BBA to health care facility (n=58) On the route to health care facility In ambulance 49 9 84.5 15.5 BBA: Birth before Arrival. Factors associated with birth before arrival Using bivariate binary logistic regression analyses, variables with a p-value of < 0.25 were recruited to be included in the final model. Thus, in the multi-variable analysis, the variables found to have an association with birth before arrival in the final model were having no antenatal care (AOR = 2.63; 95%CI: 1.23, 5.63), dependent women autonomy status (AOR = 3.32; 95%CI: 1.12, 9.89), being not knowledgeable about labor symptoms (AOR = 2.15; 95%CI: 1.11, 4.18), and having birth preparedness towards index birth (AOR = 0.13; 95%CI: 0.05, 0.35).

Therefore, this study found that women, who have no antenatal care visits during the index pregnancy, had three times higher odds of birth before arrival compared to women with antenatal care. The probability of having birth before arrival to a health care facility was three times higher for women who were dependent on their autonomy status compared with those who were autonomous. Moreover, those women who were not knowledgeable about labor symptoms had two times more likely to experience birth before arrival compared to those who were knowledgeable. Women who have birth preparedness towards index pregnancy were 87% less likely to experience birth before arrival compared to women with no birth preparedness plan. Having first and second delay, status of the road, time of delivery, and income were unrelated to the probability of birth before arrival (Table 6).

Table 6: Multivariate logistic regression showing factors associated with birth before arrival among women who gave birth in the last six months in Lemo district, Hadiya zone, Southern Ethiopia.

Variables Category COR (95% CI) AOR (95% CI) P-value Media exposure Yes No 1.00 2.09 (0.72, 6.04) 1.00 2.74 (0.82, 9.18) 0.103 Receive ANC in last pregnancy Yes No 1.00 1.77 (0.96, 3.25) 1.00 2.63 (1.23, 5.63) 0.013 Women autonomy Unautonomous Autonomous 2.19 (1.04, 4.64) 1.00 3.32 (1.12, 9.89) 1.00 0.031 Knowledge of labor symptoms Not knowledgeable Knowledgeable 2.66 (1.49, 4.75) 1.00 2.15 (1.11, 4.18) 1.00 0.023 Birth preparedness for the last birth Yes No 0.43 (0.22, 0.86) 1.00 0.13 (0.05, 0.35) 1.00 < 0.001 Used contraceptive before last pregnancy Yes No 1.31 (0.71, 2.40) 1.00 1.70 (0.78, 3.69) 1.00 0.181 First delay Delayed < 24 hours Delayed > 24 hours 1.00 1.79 (1.00, 3.24) 1.00 1.86 (0.92, 3.76) 0.082 ANC: Antenatal Care; AOR: Adjusted Odds Ratio; CI: Confidence Interval; COR: Crude Odds Ratio Discussion The prevalence of birth before arrival among women who gave birth in the last six months preceding this study in the study area was unacceptably high. In the current study, the variables associated with birth before arrival in the Lemo district of Hadiya zone were having no antenatal care, dependent women's autonomy status, being not knowledgeable about labor symptoms, and having birth preparedness towards index birth.

Globally, the prevalence of birth before arrival to a healthcare facility is estimated to be less than 1% of all deliveries in developed countries (1,5,10,14,15). But the prevalence of BBA rises exponentially in low-income countries to greater than 50% (1,7). In the current study, the prevalence of birth before arrival is 15.2%. This is a high prevalence in the study area, as the rate of BBA is used as an index of accessibility to perinatal care and a rate greater than 1.5% signals challenges in health care provision where appropriate interventions are praiseworthy (9). Births occurred between home and health care facilities either en route to health care facilities or in ambulances were given less attention and no recent evidence was found in Ethiopia that indicated its prevalence. However, according to the mini EDHS 2019 report, 40% of the total live births were delivered in health facilities in rural areas and 58.7% were delivered at home and the gap 1.2% reported as other might be taken as the prevalence of BBA to health facility even though it was not reported (7).

The current study's finding was higher than EDHS's report and this difference might be due to the misclassification bias. Accordingly, in the EDHS questionnaire, there was no option indicated for BBA, so the BBA prevalence might be misclassified to home or health facility delivery prevalence; but in the current study option for birth before arrival to health facility was indicated in the questionnaire. Yet the prevalence of BBA in South Africa is 5.4%, and in rural Malawi was 9% (4,19). As per the current study's finding, the prevalence of BBA in Lemo district was higher than the prevalence in South Africa and rural Malawi. The difference might be due to the variation of level of socio-economic status across countries.

This study established that women, who have no antenatal care visits during the index pregnancy, had three times higher odds of birth before arrival compared to women with antenatal care. Similarly, a national register study in Finland documented that one of the predictors for deliveries before arrival to health care facility was fewer prenatal visits (26). Another study from Tharaka Nithi County of Kenya documented that the obstetric risk factors associated with BBA were; ANC attendance, timing of ANC attendance and number of ANC visits (20). A prospective case control study from Nkangala District, South Africa concluded that being unbooked was found to predict the occurrence of BBAs (4). The findings of these studies were concurrent to the current study's finding. Even though there is no similar evidence from Ethiopia, our finding was supported by the 2019's mini EDHS report that showed seventy-four percent of births to mothers who attended four or more ANC visits were delivered in a health facility, as compared with 14% of births to mothers with no ANC visits (7). This signals that the ANC program if properly delivered will be important for reducing birth before arrival to health care facilities and subsequently its adverse perinatal outcomes.

Dependent women in their autonomy status compared with those who were autonomous had three times higher odds of giving birth before arrival to a health care facility as per the current study. Similarly, one study shows that women's autonomy was positively associated with health facility delivery in Ethiopia (27). Another study revealed the strongest association between delivery at healthcare facilities attended by skilled birth attendants in the Southern African region among women who made decisions on household income solely (28). Women's autonomy can influence their decision to seek health care and could result in delays in reaching as early as possible to a health care facility to give birth if she is not adequately autonomous. So this results in birth before arrival. We required policy actions that increase women's autonomy at home and this could be effective in helping assure women's delivery at health care facilites.

Furthermore, the current study reveals that those women who were not knowledgeable about labor symptoms had two times more likely to experience birth before arrival compared to those who were knowledgeable. Our finding was supported by one study from Tharaka Nithi County of Kenya which documented that the obstetric risk factors associated with BBA were recognition of the onset of labor and knowledge of signs and symptoms of labor (20). The finding implies that having poor knowledge of labor symptoms could affect women in early and properly recognizing the onset of labor and seek for healthcare facility delivery in the early hours. Therefore, standard guidelines for ANC in Ethiopia were required and emphasised that every pregnant woman should receive ANC from a skilled provider(7), which must include counselling and enter-personal education with women concerning labor symptoms.

Additionally, women who have birth preparedness towards index pregnancy were less likely to experience birth before arrival compared to women with no birth preparedness plan as per the current study. Similarly, one study from Tharaka Nithi County of Kenya documented that the obstetric risk factors associated with BBA were the identification of healthcare facility for delivery, identification of means of transport, financial preparation for hospital delivery, and basic supplies for birth (20). These are the components of the birth preparedness plan that were revealed by the Kenya study and these were used in our study as constructs to measure and compute variables for birth preparedness. As Ethiopia has adopted the WHO's goal-oriented focused antenatal care for promoting the health and survival of mothers and babies; one of its basic components that's individualized birth plan, complication readiness and emergency preparedness' is expected to alleviate the problem of BBA if properly performed. Having first and second delay, status of the raod, time of delivery, and income were unrelated to the probability of birth before arrival.

Strengths and limitations of the study Our study revealed the delivery of babies occurred between home and health care facilities and came up with the prevalence of BBA and its associated factors as this issue was given less attention by literature in Ethiopia. The study has a limitation in that it was based on a cross-sectional design due to its unclearly indicated prevalence of BBA, but we recommend it be based on a community-based case-control study. The results obtained from the current study were based on women's interviews and cannot be free from recall and social desirability biases.

Conclusion The prevalence of birth before arrival among women who gave birth in the last six months preceding this study in the study area was unacceptably high. Statistically significant association was seen between birth before arrival and having no antenatal care, dependent women autonomy status, being not knowledgeable about labor symptoms, and having birth preparedness towards index birth. Intervening to avert birth before arrival through an effective antenatal acre program especially focusing on individualized counselling concerning knowledge of labor symptoms and birth preparedness plan and providing extra vigilant attention for enhancing women's autonomy in the community may help to reduce birth before arrival and its adverse perinatal outcomes.

Data-Sharing Statement All data generated or analyzed during this study are included in the manuscript and are also available from the corresponding author upon request.

Ethical Approval and Consent to Participate Ethical clearance was obtained from Wachemo University, the faculty of medicine and the public health institution review board with reference no (WCU/NEMMCSH/182/2023). Permission was granted from the concerned bodies of Lemo woreda and selected kebele administrators. Moreover, written informed consent was obtained from each woman. Confidentiality of the information was assured. Moreover, this study was conducted in compliance with the Declaration of Helsinki. Anonymous data were taken and the confidentiality of participant's information was secured.

Acknowledgment We would like to forward our appreciations to health office and health extension workers of study area for their kind cooperation. We are also thankful to data collectors and the study participants.

Author Contributions All authors made substantial contributions to conception and design, acquisition of data, or analysis and interpretation of data; took part in drafting the article or revising it critically for important intellectual content; agreed to submit to the current journal; gave final approval of the version to be published; and agree to be accountable for all aspects of the work. All authors reviewed the manuscript.

Funding No funding was received for this work Disclosure The authors declare that they have no competing interests.

ELIGIBILITY:
Postpartum women who were in a state of not being able to respond to the study questionnaires due to their health status were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: A community-based cross-sectional study was conducted among 382 postpartum women who gave birth in the last six months before the current study and reside in Lemo Woredas.
Sampling Method: Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Birth before Arrival | May, 2023

SECONDARY OUTCOMES:
Associated Factors of Birth Before Arrival among Postpartum Women | May, 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Wachemo University, Hosa’ina, Ethiopia

IPD SHARING:
Plan to Share IPD: No